CLINICAL TRIAL: NCT05153876
Title: NLP Headache Open: an Open Internet-based Survey and Natural Language Processing Project Analysing Written Monologues by Headache Patients
Brief Title: An Open Internet-based Survey and Natural Language Processing Project Analysing Written Monologues by Headache Patients
Acronym: NLPH-OPEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10635
Record Dates: First submitted 2021-10-01; First posted 2021-12-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Headache Disorders; Tension-Type Headache; Migraine Disorders; Cluster Headache; TACS; Secondary Headache Disorder
Keywords: Migraine; Natural Language Processing; Headache
MeSH Terms: conditions — Headache Disorders; Tension-Type Headache; Migraine Disorders; Cluster Headache; Headache Disorders, Secondary; Headache | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants filling in the questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Headache attack descriptions, Headache related disability descriptions, Questionnaires, MIDAS, MSQv2.1, SF36

SUMMARY:
Headache disorders are among the most prevalent medical conditions worldwide. The diagnosis of headache disorders is based on medical history taking. Digital solutions such as natural language processing (NLP) may be of aid to understand the linguistic aspects of headache attack and headache related disability descriptions by patients. Participants will provide a written description of their headache disorder. The results will hopefully lead to a better understanding of the potential use of NLP in headache disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* Have a headache disorder with at least one headache attack over the last three months
* voluntary participation
* accepted the patient information sheet and gave informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with headache disorders
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Lexical diversity and differences between migraine and cluster headache | through study completion, an average of 1 year
  Chi-square measurement of a word token used by migraine patients versus cluster headache patients

SECONDARY OUTCOMES:
Accuracy of machine learning experiments for the correct classification of headache disorders | through study completion, an average of 1 year
  Machine learning experiments to investigate the potential to build modelling algorithms that accurately classify the self-given diagnosis by the patient based on text.
F1 scores of machine learning experiments for the correct classification of headache disorders | through study completion, an average of 1 year
  Machine learning experiments to investigate the potential to build modelling algorithms that accurately classify the self-given diagnosis by the patient based on text.
Word counts | through study completion, an average of 1 year
  Counts of word tokens of different headache disorder groups
Sentences counts | through study completion, an average of 1 year
  Counts of sentence tokens of different headache disorder groups
Paragraph counts | through study completion, an average of 1 year
  Counts of paragraph tokens of different headache disorder groups
Term-frequency inverse document frequency scores (TF-IDF) | through study completion, an average of 1 year
  TF-IDF scores of word tokens of different headache disorder groups
Migraine Disabillity Assessment [MIDAS] score calculation with text input | through study completion, an average of 1 year
  Machine learning experiments to investigate the potential to build modelling algorithms that accurately predict the impact score from Migraine Disabillity Assessment [MIDAS] based on text.
Migraine Specific Questionaire versie 2.1 [MSQv2.1] score calculation with text input | through study completion, an average of 1 year
  Machine learning experiments to investigate the potential to build modelling algorithms that accurately predict the impact score from Migraine Specific Questionaire versie 2.1 [MSQv2.1] based on text.
RAND SF-36 Dutch version score calculation with text input | through study completion, an average of 1 year
  Machine learning experiments to investigate the potential to build modelling algorithms that accurately predict the impact score from RAND SF-36 Dutch version based on text.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent: Department of Neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No